CLINICAL TRIAL: NCT04446351
Title: A Phase 1 First-Time-in-Human, Open-Label Study of GSK6097608 Administered as Monotherapy and in Combination With Anticancer Agents in Participants With Advanced Solid Tumors
Brief Title: Study of the Safety and Effectiveness of GSK6097608 in Participants With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: 23andMe, Inc. (Industry); iTeos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 212214
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Neoplasms
Keywords: GSK6097608; dostarlimab; Dose escalation; Pharmacokinetics; Pharmacodynamics; Advanced solid tumors; First-time-in-human; GSK4428859A; EOS884448; cobolimab; belrestotug
MeSH Terms: conditions — Neoplasms | interventions — dostarlimab

STUDY DESIGN:
Intervention Model Description: Participants will receive treatment in different dose escalation arms of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Participants receiving GSK6097608 monotherapy (Arm A) (Experimental): Participants will be administered an intravenous (IV) infusion of GSK6097608 every 3 weeks as monotherapy in escalating doses.
  Interventions: Drug: GSK6097608
- Participants receiving GSK6097608 plus dostarlimab (Arm B) (Experimental): Participants will be administered IV infusion of GSK6097608 every 3 weeks in escalating doses followed by dostarlimab.
  Interventions: Drug: GSK6097608; Drug: Dostarlimab
- Participants receiving dostarlimab monotherapy (Arm D) (Experimental): Participants will be administered an IV infusion of dostarlimab monotherapy (1 cohort will receive dostarlimab every 3 weeks and 1 cohort will receive dostarlimab every 6 weeks).
  Interventions: Drug: Dostarlimab
- Participants receiving dostarlimab plus belrestotug (Arm E) (Experimental): Participants will be administered IV infusions of dostarlimab followed by belrestotug, every 3 weeks.
  Interventions: Drug: Dostarlimab; Drug: Belrestotug
- Participants receiving dostarlimab plus belrestotug plus GSK6097608 (Arm F) (Experimental): Participants will be administered an IV infusion of dostarlimab followed by belrestotug followed by GSK6097608 every 3 weeks.
  Interventions: Drug: GSK6097608; Drug: Dostarlimab; Drug: Belrestotug
- Participants receiving dostarlimab plus cobolimab (Arm G) (Experimental): Participants will be administered an IV infusion of cobolimab followed by dostarlimab
  Interventions: Drug: Dostarlimab; Drug: Cobolimab

INTERVENTIONS:
Drug: GSK6097608 — GSK6097608 will be administered as an IV infusion.
  Arms: Participants receiving GSK6097608 monotherapy (Arm A); Participants receiving GSK6097608 plus dostarlimab (Arm B); Participants receiving dostarlimab plus belrestotug plus GSK6097608 (Arm F)
Drug: Dostarlimab — Dostarlimab will be administered as an IV infusion.
  Arms: Participants receiving GSK6097608 plus dostarlimab (Arm B); Participants receiving dostarlimab monotherapy (Arm D); Participants receiving dostarlimab plus belrestotug (Arm E); Participants receiving dostarlimab plus belrestotug plus GSK6097608 (Arm F); Participants receiving dostarlimab plus cobolimab (Arm G)
Drug: Cobolimab — Cobolimab will be administered as an IV infusion.
  Arms: Participants receiving dostarlimab plus cobolimab (Arm G)
Drug: Belrestotug — Belrestotug will be administered as an IV infusion.
  Other Names: GSK4428859A; EOS884448
  Arms: Participants receiving dostarlimab plus belrestotug (Arm E); Participants receiving dostarlimab plus belrestotug plus GSK6097608 (Arm F)

SUMMARY:
This first-time-in-human (FTIH) study will evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary clinical activity of escalating doses of GSK6097608 given as monotherapy and in combination with dostarlimab in participants with advanced solid tumors. In addition, dostarlimab will be given as monotherapy (Arm D); and in combination with belrestotug (Arm E); and with GSK6097608 + belrestotug (Arm F) in Japanese and Chinese participants. The study may assess the PK/PD cohorts for Arm E and/or Arm F in participants outside of China and Japan. Additionally, dostarlimab will be given in combination with cobolimab in Japanese participants. Drug name mentioned as belrestotug, GSK4428859A and EOS884448 are interchangeable for the same compound. In the rest of the document, the drug will be referred to as belrestotug.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older (or >=20 years of age in Arm-A Japan, Arm-D Japan, Arm E-Japan, Arm F-Japan, and Arm G-Japan)
* Female participants of childbearing potential must agree to use a highly effective form of contraception
* Histological or cytological documentation of locally advanced, recurrent, or metastatic solid malignancy. Enrollment in PK/PD cohorts will be restricted to participants with histologically or cytologically confirmed diagnosis of 1 or more of the following: non-small-cell lung cancer (NSCLC), head and neck squamous cell carcinoma (HNSCC), endometrial cancer (EC), colorectal cancer (CRC) (including specified molecular subtypes of these) or an alternative immunogenic tumor type with medical monitor approval
* Disease that has progressed after standard therapy for the specific tumor type, or for which standard therapy has proven to be ineffective, intolerable, or is considered inappropriate, or if no further standard therapy exists
* Participants in a PK/PD cohort (Arms A, B, E and F) must provide fresh tumor biopsies. Biopsies are not required from participants enrolled in Arm D, Arm E, (non-PK/PD cohorts only), Arm F (non-PK/PD cohort only), Arm G or any participant enrolled in mainland China
* Eastern cooperative oncology group (ECOG) performance status (PS) 0 to 1
* Life expectancy of at least 12 weeks
* Adequate organ function as determined by laboratory assessments
* Adequate cardiac ejection fraction as measured by echocardiogram
* Arm A-Japan, Arm D-Japan, Arm E-Japan, Arm F-Japan, and Arm G-Japan only: lives in Japan and is racially Japanese, defined as all biological grandparents being Japanese
* Arm A-China, Arm B-China, Arm D-China, Arm E-China and Arm F-China only (excluding PK/PD cohorts in Arm E and Arm F): is of Chinese descent and lives in China
* Arm D, Arm E, Arm F, and Arm G only: has been deemed suitable for assigned treatment based on assessment by the investigator

Exclusion Criteria:

* Prior anti-cancer treatment including investigational agents, immune checkpoint inhibitors, chemotherapy, targeted therapy, and biological therapy: within 4 weeks or 5 half-lives of the drug, whichever is shorter
* Prior allogenic or autologous bone marrow transplantation or other solid organ transplantation
* Toxicity from previous anticancer treatment, including; greater than or equal to (>=) Grade 3 immune-mediated toxicity considered related to prior immunotherapy and that led to treatment discontinuation; or toxicity related to prior treatment that has not resolved; or history of myocarditis of any grade during a previous treatment with immunotherapy
* Known additional malignancy that progressed or required active treatment within the last 2 years
* Uncontrolled or symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis
* Active autoimmune disease that has required systemic disease-modifying or immunosuppressive treatment within the last 2 years
* Concurrent medical condition requiring the use of systemic immunosuppressive treatment
* Cirrhosis or current unstable liver or biliary disease per investigator assessment
* Active infection requiring systemic treatment, known human immunodeficiency virus infection, or positive test for hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV)
* Prolonged QT as measured by electrocardiogram
* Allergen desensitization therapy within 4 weeks of starting study intervention
* History of hypersensitivity to any of the study interventions or their excipients
* Has a history or evidence of cardiac abnormalities within the 6 months prior to enrolment
* Recent history (within 6 months) of uncontrolled symptomatic ascites or pleural effusions
* History of idiopathic pulmonary fibrosis; interstitial lung disease; organizing pneumonia; noninfectious pneumonitis that required steroids, or evidence of active, noninfectious pneumonitis
* Pregnant or lactating woman
* Receipt of live vaccine within 30 days of the start of study intervention
* Receipt of transfusion of blood products or administration of colony-stimulating factors within 14 days before the first dose of study intervention
* Major surgery less than 4 weeks before the first dose of study intervention
* Known drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicities (DLTs) | Up to Day 21
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to 2 years

SECONDARY OUTCOMES:
Number of participants with clinically significant changes in laboratory parameters, vital signs, and 12-lead electrocardiogram (ECG) findings | Up to 2 years
Number of participants with dose reductions or delay | Up to 2 years
Number of participants withdrawn due to AEs | Up to 2 years
Overall response rate (ORR) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | Up to 2 years
Arms D, E, F, G: ORR based on modified Response Evaluation Criteria in Solid Tumors (iRECIST) | Up to 2 years
Arms D, E, F, G: Disease Control Rate (DCR) based on RECIST 1.1 | Up to 2 years
Arms D, E, F, G: DCR based on iRECIST | Up to 2 years
Arms D, E, F, G: Time to response (TTR) based on RECIST 1.1 | Up to 2 years
Arms D, E, F, G: TTR based on iRECIST | Up to 2 years
Arms D, E, F, G: Duration of response (DOR) based on RECIST 1.1 | Up to 2 years
Arms D, E, F, G: DOR based on iRECIST | Up to 2 years
Arms D, E, F, G: Progression-free survival (PFS) based on RECIST 1.1 | Up to 2 years
Arms D, E, F, G: PFS based on iRECIST | Up to 2 years
Arms A, B, F: Number of participants with positive anti-drug antibodies (ADAs) against GSK6097608 | Up to 2 years
Arms A, B, F: Titers of ADAs against GSK6097608 | Up to 2 years
Arms B, D, E, F, G: Number of participants with positive ADAs against dostarlimab | Up to 2 years
Arms B, D, E, F, G: Titers of ADAs against dostarlimab | Up to 2 years
Arms E, F: Number of participants with positive ADAs against belrestotug | Up to 2 years
Arms E, F: Titers of ADAs against belrestotug | Up to 2 years
Arm G: Number of participants with positive ADAs against cobolimab | Up to 2 years
Arm G: Titers of ADAs against cobolimab | Up to 2 years
Arms A, B, F: Maximum observed concentration (Cmax) for GSK6097608 | Up to 2 years
Arms A, B, F: Minimum observed concentration (Cmin) for GSK6097608 | Up to 2 years
Arms A, B, F: Area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC[0-infinity]) for GSK6097608 | Up to 2 years
Arms A, B, F: Area under the plasma concentration-time curve from time zero to time (AUC[0-t]) for GSK6097608 | Up to 2 years
Arms A, B, F: Apparent terminal phase half-life (t1/2) for GSK6097608 | Up to 2 years
Arms B, D, E, F, G: Cmax for dostarlimab | Up to 2 years
Arms B, D, E, F, G: Cmin for dostarlimab | Up to 2 years
Arms B, D, E, F, G: AUC(0-infinity) for dostarlimab | Up to 2 years
Arms B, D, E, F, G: AUC(0-t) for dostarlimab | Up to 2 years
Arms B, D, E, F, G: t1/2 for dostarlimab | Up to 2 years
Arms E, F: Cmax for belrestotug | Up to 2 years
Arms E, F: Cmin for belrestotug | Up to 2 years
Arms E, F: AUC(0-infinity) for belrestotug | Up to 2 years
Arms E, F: AUC(0-t) for belrestotug | Up to 2 years
Arms E, F: t1/2 for belrestotug | Up to 2 years
Arm G: Cmax for cobolimab | Up to 2 years
Arm G: Cmin for cobolimab | Up to 2 years
Arm G: AUC(0-infinity) for cobolimab | Up to 2 years
Arm G: AUC(0-t) for cobolimab | Up to 2 years
Arm G: t1/2 for cobolimab | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- United States (5):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
- Canada (2):
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
- Japan (2):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/